CLINICAL TRIAL: NCT04492852
Title: Comparison of Surgical Site Infection After Skin Closure by Prolene or Staples in Bilateral Knee Arthroplasty Patients: A Parallel Design Randomized Controlled Trial
Brief Title: Comparison of Surgical Site Infection After Skin Closure by Prolene or Staples in Bilateral Knee Arthroplasty Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indus Hospital and Health Network (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ahsun Jiwani, Junior Biostatistician, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 456-784-7
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Total Knee Replacement
Keywords: Knee Replacement; Prolene; Staples; Surgical Site Infection; Skin Closure
MeSH Terms: conditions — Surgical Wound Infection | interventions — Polypropylenes; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm 1 (Experimental): After total knee replacement, the skin closure of the patients in this group will be done using polypropylene (PROLENE) sutures.
  Interventions: Procedure: Polypropylene (PROLENE) sutures
- Interventional Arm 2 (Active Comparator): After total knee replacement, the skin closure of the patients in this group will be done using staple sutures.
  Interventions: Procedure: Staple Sutures

INTERVENTIONS:
Procedure: Polypropylene (PROLENE) sutures — After total knee replacement, the skin closure of the patients in this group will be done using polypropylene (PROLENE) sutures.
  Arms: Interventional Arm 1
Procedure: Staple Sutures — After total knee replacement, the skin closure of the patients in this group will be done using staple sutures.
  Arms: Interventional Arm 2

SUMMARY:
Knee arthroplasty also known as the total knee replacement is an orthopedic surgical procedure done to resurface the knee that has been severely damaged by arthritis. The optimal goal of skin closure after the procedure is to promote rapid healing and an acceptable cosmetic result while minimizing the risk of infection. Skin closure after knee arthroplasty is done by using either of the two widely used sutures i.e. polypropylene (Prolene) sutures or the skin staple sutures. The literature is very scarce on knee arthroplasty patients and the results of the studies conducted have been inconclusive of the studies conducted on the patients of knee arthroplasty. Moreover, there are no standard guidelines as to which type of suture should be used. The type of sutures is being selected on the orders and wishes of the surgeon at the time of skin closure. Prolene sutures are made up of a synthetic steroisomer known as polypropylene. It is a monofilament non-absorbable, sterile surgical suture. They are indicated for use in general soft tissue. It Provides permanent tensile strength retention in tissue, even in the presence of infection. These sutures are exceptionally smooth for an easy passage through the tissue. Prolene sutures are widely used in cardiovascular, orthopedics, ophthalmic, and neurological surgical procedures. Another type of sutures that are used to close the surgical wound are the staple sutures. They are used as an alternative to the traditional Prolene sutures. They are non-absorbable and usually used on surgical wounds that are big, complex or hard to close by using Prolene. These are specialized staples made up of titanium, stainless steel or plastic.

Interventions:

The study will have 2 intervention arms. The patients will be randomized to receive either Prolene sutures for wound closure or staple sutures for wound closure. After the application of the intervention, routine care would be given to the patients postoperatively.

Hypothesis:

The investigators hypothesize that there is no difference in the incidence of surgical site infection in bilateral TKR patients with wound closure by Prolene vs staple.

Study Design:

This study will be conducted as an open blinded, parallel design, equivalence randomized controlled trial. The patients would be randomized to receive either of the two interventions i.e. Prolene or Staple sutures.

DETAILED DESCRIPTION:
Study Enrollment Procedures:

Enrollment will be a continuous process with screening and enrolling eligible patients admitted through the clinic electively for primary TKR. Informed consent will be taken from the patient as per routine protocol before the arthroplasty procedures in the hospital. Research objectives, methodology, risks, and benefits will be explained in detail. Consent for the participation in the study will only be taken by the primary investigator at his clinic or the surgical resident on call preoperatively along with the consent for the surgical procedure.

Pre-Randomization Evaluations Screening:

The screening will involve the routine history taking and physical examination by the doctor and nursing staff in the clinic. Screening won't involve performing procedures that are not part of routine management.

On-study/on-intervention evaluations:

After screening and assessing the eligibility, patients will be randomly allocated by a 1:1 ratio to the two intervention groups i.e. prolene or staple using a computer-generated randomization sequence by the clinical trials unit (CTU), which they will provide to the PI, after patients' admission in the hospital. Patients will be followed from the time they reach the ward after surgery until their hospital discharge, which is usually around 7 days.

Data Collection:

The data collection will be done by the surgical site infection (SSI) nurses from the infection control department of AKUH. These nurses are well-trained to assess the surgical site infections in all the surgery patients admitted to the hospital. Training of data collectors will be done by the PI to ensure the reliability and validity of the study. The data collectors will be strictly instructed to respect the autonomy of participants. Data collection will be done by the data collectors under the supervision of the PI and CTU. Questionnaires will be checked for consistency and logical data entries. Data entry will be done, and counter checked by the PI at regular intervals.

Data Storage:

Data collected will be coded and kept confidential without the identifiable information of patients. The confidentiality of the study participants will be maintained throughout the study period. Data collected will be kept confidential without identifiable information of patients who are identified by a number assigned. The hard copy forms will be retained in a secured location with the PI after data entry into computer software and will be kept as per hospital protocol. The password-protected drives will be used to store data with only the PI having access to it. The data will be available for AKUH ethical review committee on request and might be published in a journal without disclosing any identifiable information of patients. Filled questionnaires will be stored for 5 years after the study is completed as per the policy of the institute.

Sample Size:

The sample size was calculated via open epi software version 3.01. The level of significance was kept at 5% with a power of 80%. The percentage of exposed (staple sutures) with outcome (surgical site infection) was 66%. The percentage of non-exposed (Prolene sutures) with outcome (surgical site infection) was 33%. The estimated risk ratio taken from a study was 2. After adding the non-response rate of 10% the final sample size came out to be 82 patients with 41 patients in each arm.

Plan of Analysis:

Statistical analysis will be done by using STATA software version 15. The normality assumption for the quantitative variables would be assessed using the shapiro wilk test. Mean ± SD will be computed for all the normally distributed quantitative variables. The median and interquartile range would be reported for the non-normally distributed quantitative variables. The categorical variables would be expressed in frequencies and percentages. The Cox Proportional Hazard regression will be used for the univariate and multivariable analysis. Univariate analysis will be conducted, and crude risk ratios and their 95% confidence intervals will be obtained. All significant independent variables at the univariate stage will be regressed in a multivariable cox proportional hazard regression using the stepwise method in the multivariable model and the adjusted risk ratios will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of age 40-70 years
* Undergoing bilateral knee arthroplasty at AKUH Karachi.
* Both the genders would be included.
* Patients having American Society of Anesthesiologists (ASA) level of I, II and III
* Patients having functional class of I, II and III pre-operatively
* Patients opting to undergo Bilateral knee arthroplasty under care of the selected surgeon (A) for the study.
* Patients undergoing bilateral TKR electively

Exclusion Criteria:

* Patients unwilling to consent.
* Patients unable to comprehend due to the language barrier
* Patients who have a Glasgow Coma Scale i.e. GCS<15 (cognitive impairment)
* Patients undergoing a knee revision surgery
* Patients having a previous incision/scar in the operative field will be excluded
* Patients having documented allergy to Prolene or stainless steel
* Patients having a documented underlying malignancy
* Patients undergoing unilateral TKR or staged bilateral TKR
* Patients undergoing emergency TKR.
* Patients having undergoing surgery due to trauma or fracture

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 6 weeks for superficial infections and 1 year for deep infections
  Primary outcome of the study is the incidence of surgical site infection (superficial or deep) within 6 weeks for superficial infections and 1 year for deep infections.

SECONDARY OUTCOMES:
Post Operative complications | Within 2 weeks of surgery
  The secondary outcomes of the study include the incidence of post-operative complication that includes; seroma, hematoma, pain, or bleeding
Pain Score | post-operative follow up at 14th post-op day
  assess and compare the pain scores at the time of suture removal using the Visual Analogue Scale (VAS) pain scale. score of '0' represents no pain whereas a score of '10' represents severe/unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsun Jiwani, MSc. Epibio, Principal Investigator — The Indus Hospital

REFERENCES:
- [Background] Liu S, Wang Y, Kotian RN, Li H, Mi Y, Zhang Y, He X. Comparison of Nonabsorbable and Absorbable Suture in Total Knee Arthroplasty. Med Sci Monit. 2018 Oct 23;24:7563-7569. doi: 10.12659/MSM.910785. PMID 30350827
- [Background] Barrow J, Divecha H, Board T. Skin closure in arthroplasty surgery: Current practice. Int Wound J. 2018 Dec;15(6):966-970. doi: 10.1111/iwj.12956. Epub 2018 Jul 6. PMID 29978557
- [Result] Smith TO, Sexton D, Mann C, Donell S. Sutures versus staples for skin closure in orthopaedic surgery: meta-analysis. BMJ. 2010 Mar 16;340:c1199. doi: 10.1136/bmj.c1199. PMID 20234041
- [Result] Gatt D, Quick CR, Owen-Smith MS. Staples for wound closure: a controlled trial. Ann R Coll Surg Engl. 1985 Sep;67(5):318-20. PMID 3901864
- [Result] Clayer M, Southwood RT. Comparative study of skin closure in hip surgery. Aust N Z J Surg. 1991 May;61(5):363-5. doi: 10.1111/j.1445-2197.1991.tb00235.x. PMID 2025190
- [Result] Khan RJ, Fick D, Yao F, Tang K, Hurworth M, Nivbrant B, Wood D. A comparison of three methods of wound closure following arthroplasty: a prospective, randomised, controlled trial. J Bone Joint Surg Br. 2006 Feb;88(2):238-42. doi: 10.1302/0301-620X.88B2.16923. PMID 16434531
- [Derived] Hasan O, Jiwani A, Mazhar L, Begum D, Lakdawala R, Noordin S. Comparison of Surgical Site Infection After Skin Closure by Prolene or Staples in Bilateral Simultaneous Knee Arthroplasty Patients: A Parallel Design Randomized Controlled Trial Protocol. Int J Surg Protoc. 2021 Aug 6;25(1):154-159. doi: 10.29337/ijsp.153. eCollection 2021. PMID 34430763